CLINICAL TRIAL: NCT04475796
Title: Early Versus Delayed Laparoscopic Cholecystectomy Following ERCP in Concomitant Gallstones and Common Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Aouf, Dr, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 124569124569
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Choledocholithiasis With Cholecystitis
Keywords: Choledocholithiasis; Early; Delayed; Laparoscopic cholecystectomy; ERCP; Nassar scale
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early group (Active Comparator)
  Interventions: Procedure: Laparoscopic cholecystectomy
- Delayed group (Active Comparator)
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy performed after ERCP

SUMMARY:
The present study aimed to compare early and delayed laparoscopic cholecystectomy after ERCP for CBDs and gallstones.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) followed by laparoscopic cholecystectomy (LC) is a commonly performed treatment modality for concomitant common bile duct stones (CBDs) and gallbladder stones. There has been a debate about the appropriate timing of laparoscopic cholecystectomy after ERCP. The present study aimed to compare early and delayed laparoscopic cholecystectomy after ERCP for CBDs and gallstones adding new parameters like Nassar scale.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopic cholecystectomy after clearance of CBDs by ERCP

Exclusion Criteria:

* advanced liver cirrhosis, pancreatitis, acute cholangitis, suspected malignancy, severe malnutrition, and pregnancy.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — adult
Enrollment: 66 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
operative time | one day
  the time to perform laparoscopic cholecystectomy from the time of incision to the last suture

SECONDARY OUTCOMES:
intraoperative difficulty and complications | one day
  the difficulties that face the surgeon during the surgery and the early complications that result

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aouf, Dr., Principal Investigator — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt